CLINICAL TRIAL: NCT02907502
Title: Effects of Milk Protein Intake in Young Children on Early Growth and Later Obesity Risk: a Multicentre Randomized Clinical Trial
Brief Title: Toddler Milk Intervention Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 13.29.INF
Record Dates: First submitted 2016-08-31; First posted 2016-09-20 (Estimated); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental formula (Experimental): Young-child formula with low protein content
  Interventions: Dietary Supplement: Young-child formula with low protein content
- Control formula (Active Comparator): Young-child formula with protein content similar to that of cow's milk
  Interventions: Dietary Supplement: Young-child formula with protein content similar to that of cow's milk

INTERVENTIONS:
Dietary Supplement: Young-child formula with low protein content — Young-child formula with low protein content
  Arms: Experimental formula
Dietary Supplement: Young-child formula with protein content similar to that of cow's milk — Young-child formula with protein content similar to that of cow's milk
  Arms: Control formula

SUMMARY:
To assess growth of children (enrolled between 11.5 and 13.5 months) fed with two iso-energetic, young-child formulas with different protein content during the second year of life

DETAILED DESCRIPTION:
This study is designed to investigate in a randomized double-blind parallel-group trial the growth and metabolic effects of different contributions of protein to total energy intakes in healthy children during the second year of life

ELIGIBILITY:
Inclusion Criteria:

* Having obtained his/her parents' (or his/her legally accepted representative [LAR's] written informed consent and having evidence of personally signed and dated informed consent document indicating that the child's parents/LAR have been informed of all pertinent aspects of the study
* Child was born full term (≥ 37 weeks of gestation)
* Age at enrollment: between 11.5 months and 13.5 months of age
* 2.5 kg ≤ birth weight ≤ 4.5 kg
* Born from a singleton pregnancy
* Child's parent(s)/LAR is of legal age of consent, has sufficient local language skills to complete the informed consent and other study documents, is able to be contacted directly by telephone throughout the study, and is willing and able to fulfill the requirements of the study protocol.

Exclusion Criteria:

* Diagnosed disorder considered to interfere with nutrition or growth (e.g. malabsorptive disorders as short bowel syndrome, inflammatory bowel disease; neurological and congenital disorders that may delay growth as cerebral palsy, agenesis of the corpus callosum, spina bifida, Down Syndrome, Cri Du Chat; disorders that may lead to obesity: Prader willi syndrome, Angelman syndrome, etc.)
* Cows' milk allergy
* Lactose intolerance
* Participation in any other interventional clinical trial during the 4 weeks prior to enrollment
* Infant who is being breastfed at the time of enrollment
* Infant who does not usually drink 300ml of cow's and/or formula milk per day
* Institutionalized children
* Child or child's family who in the Investigator's judgment cannot be expected to comply with the protocol or study procedures

Ages: 11 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1618 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2024-10 (Actual)

PRIMARY OUTCOMES:
BMI-for-age z-score | Age 24 months
  WHO-growth standard

SECONDARY OUTCOMES:
BMI-for-age z-score | Age 72 months
The percentage of overweight and obese children | Age 24 months
  CDC definition: Overweight above 85th to less than the 95th percentile and obese 95th percentile or greater and analyzed by the method of Peacock (Dichotomising continuous data while retaining statistical power using a distributional approach, Statistics in medicine, 2012).
The percentage of overweight and obese children | Age 72 months
Growth parameters: Anthropometry: Weight, Length, Heel knee length, Mid-arm circumference, Waist circumference, Hip circumference (only 48 months and 72 months), Head circumference, Triceps skinfold, Subscapular skinfold | Age 12, 18, 24, 48 and 72 months
Child's development: Parental rating of child development with Ages & Stages Questionnaires® | Age 24 and 48 months
Body composition: air displacement plethysmography | at 24, 48 and 72 months of age
Metabolomic profile: Plasma and urine metabolic indicators of energy and protein metabolism (metabolomics with a focus on carnitines, amino acid catabolism, ketone bodies, Krebs cycle, and bacterial utilization of protein and carbohydrates) | Age 12, 18, 24, 48 and 72 months
DNA methylation pattern: Methylation status of specific DNA regions (e.g. CpG sites) | Age 12, 24 and 72 months
Blood pressure | Age 48 and 72 months
Dietary intake: 24-hour recall | Age 12, 18, 24, 48 and 72 months
Metabolic and endocrine markers: Blood and Urine markers | Age 12, 24 and 72 months
  Blood: Complete blood count, Glucose, Creatinine, Ferritin (measured only at 24 months), 25-OH vitamin D (measured only at 24 months), Triglycerides, Total cholesterol, HDL- and LDL-cholesterol, Insulin, FGF-21, IGF-1, IGF-BP2, IGF-BP3, Leptin, Adiponectin, Ghrelin, Amino Acids, Serum albumin, Urea, C-reactive protein, Osteocalcin / Urine: Calcium, C-peptide, Creatinine, Urea nitrogen

CONTACTS AND LOCATIONS:
Locations (2):
- Dr Von Hauner Children's hospital, Munich, Germany
- Hospital Universitari Joan 23 de Tarragona. Universitat Rovira i Virgili., Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neiss J, Demmelmair H, Geyer F, Triebswetter A, Angkasa D, Escribano J, Ferre N, Gispert-Llaurado M, Koletzko B, Bechtold-Dalla Pozza S, Grote V. Associations of insulin-like growth factor 1 and IGF binding proteins 2 and 3 with lipids in toddlers. Lipids Health Dis. 2026 Feb 3. doi: 10.1186/s12944-026-02872-y. Online ahead of print. PMID 41634786
- [Derived] Ferry JM, Escribano J, Gispert-LLaurado M, Koletzko B, Grote V. Impact of cut-point methods on classification of physical activity and sedentary behaviour of toddlers. BMC Public Health. 2025 Oct 2;25(1):3290. doi: 10.1186/s12889-025-24636-6. PMID 41039386
- [Derived] Grote V, Jaeger V, Escribano J, Zaragoza M, Gispert M, Grathwohl D, Koletzko B. Effect of milk protein content in Toddler formula on later BMI and obesity risk: protocol of the multicentre randomised controlled Toddler Milk Intervention (ToMI) trial. BMJ Open. 2021 Dec 7;11(12):e048290. doi: 10.1136/bmjopen-2020-048290. PMID 34876419